CLINICAL TRIAL: NCT06218316
Title: Combined Effect of Repetitive Transcranial Magnetic Stimulation and Botulinum Injection on Spasticity and Motor Functions of Children With Diplegic Cerebral Palsy
Brief Title: Repetitive Transcranial Magnetic Stimulation Versus Botulinum Injection on Spasticity on Children With Diplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Rana Nabil Hussein Mohamed, lecturer of pediatric physical therapy, MTI University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004846
Record Dates: First submitted 2023-12-28; First posted 2024-01-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Spastic Diplegic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A; Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: one-way analysis of variance (ANOVA)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Botox for spasticity (Experimental): Botox for spasticity in lower limbs in cerebral palsy children
  Interventions: Drug: botulinum toxin A; Other: Rehabilitation Training Protocol
- transcranial magnetic stimulation for spasticity (Experimental): transcranial magnetic stimulation for spasticity in cerebral palsy children
  Interventions: Device: Transcranial Magnetic Stimulation; Other: Rehabilitation Training Protocol
- Botox combined with transcranial magnetic stimulation for spasticity (Experimental): Botox combined with transcranial magnetic stimulation for spasticity in cerebral palsy children
  Interventions: Drug: botulinum toxin A; Device: Transcranial Magnetic Stimulation; Other: Rehabilitation Training Protocol

INTERVENTIONS:
Drug: botulinum toxin A — Botulinum Neurotoxin A (BoNT-A) Injections will administered directly into the bulk of the muscles, with two injection sites at each head of the gastrocnemius and two sites into the medial hamstring. one vial of BoNT-A in 2 mL of 0.9% sodium chloride solution. followed by a 3-month rehabilitation program. The entire intervention including rTMS, BoNT-A, and rehabilitation training program spanned a period of three months.
  Arms: Botox combined with transcranial magnetic stimulation for spasticity; Botox for spasticity
Device: Transcranial Magnetic Stimulation — Repeated Transcranial Magnetic Stimulation (rTMS) Stimulation coil will strategically place on the primary motor cortex (M1), The patients received 1500 pulses per session, two sessions per week for 3 months, in a combination with 3-month rehabilitation program.
  Arms: Botox combined with transcranial magnetic stimulation for spasticity; transcranial magnetic stimulation for spasticity
Other: Rehabilitation Training Protocol — Rehabilitation Training Protocol: As part of the study protocol, all participating children underwent a comprehensive weekly routine rehabilitation training program. Training Schedule: sessions will conduct for duration of 45 minutes. Training occurred four days a week.

SUMMARY:
This trial will enroll 75 children with spastic diplegic cerebral palsy both matched in age, sex, degree of disability and cognitive functions with the same exclusion criteria undergoing the same physical therapy. All enrolled children will undergo routine physical therapy program and will be divided into three groups (n = 25 per group) according treatment methods. Group A: children will be given local injections of botulinum toxin type ,Group B: children will be given repetitive transcranial magnetic stimulation on the affected side; Group C: children will be given local injections of botulinum toxin type A combined with repetitive transcranial magnetic stimulation , the three groups will take physical therapy (PT) of 45 minutes duration 4 days a week for 3 months .The grade of spasticity will be assessed by using Modified Ashworth scale and M/H ratio by using EMG. The grade of motor function will assessed by using Gross Motor Function Classification System (GMFCS).

DETAILED DESCRIPTION:
This trial will enrol 75 children with spastic diaplegic cerebral palsy with both sex, degree of disability and cognitive functions with the same exclusion criteria and the same physical therapy program. All enrolled children will undergo routine physical therapy program and will be divided into three groups (n = 25 per group) according treatment methods. Group A: children will be given local injections of botulinum toxin type ,Group B: children will be given repetitive transcranial magnetic stimulation on the affected side; Group C: children will be given local injections of botulinum toxin type A combined with repetitive transcranial magnetic stimulation , the three groups will take physical therapy (PT) of 45 minutes duration 4 days a week for 3 months.

They will diagnosed based on history taking including perinatal, developmental, and family history, general and neurological examination. The included children with clinical diagnosis of moderate spastic diplegic cerebral palsy with a MAS (1, 1+, 2) and GMFCS (II, III, IV) will participated in this study. On the contrary, children with dyskinetic CP, mental retardation, previous ankle or knee surgery, uncontrolled epileptic seizure or contracture will excluded

ELIGIBILITY:
Inclusion Criteria:

* were diagnosed based on history taking including perinatal, developmental, and family history, general and neurological examination.

The included children with clinical diagnosis of moderate spastic dialogic cerebral palsy with a MAS (1, 1+, 2) and GMFCS (II, III, IV) were participated in this study

Exclusion Criteria:

Children who's contraindicated to rTMS treatment have metal implants such as internal pacemakers and intracranial scaffolds, and/or a history of epilepsy.

* Children who's Contraindicated for BTX-A treatment: hypersensitivity and local infection at the injection site.
* Children which have received a local injection of BTX-A within 3 months.
* Children with dyskinetic CP,
* Mental retardation,
* previous, seizure or contracture were excluded.

Ages: 4 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
modified aswthor scale | 3 months
  Modified Ashworth Scale (MAS): The MAS measures the resistance and spasticity in the joint during passive movement. The resistance is scored from 0 to 5 (0 the least severe to 5 the most severe

SECONDARY OUTCOMES:
Gross Motor Function Classification System | 3 months
  Gross Motor Function Classification System (GMFCS): The GMFCS provides a standardized system to classify the gross motor function of children with CP into five levels (level I the least severe to level V the most severe)

OTHER OUTCOMES:
Electromyography | 3 months
  The Hofmann's reflex or H-reflex, as measured by electromyography (EMG), has been used to assess spasticity. The H-reflex measures the threshold spinal reflex reaction in muscles after electrical stimulation of the peripheral nerve, believed to be indicative of alpha motor neuron excitability. People with spasticity have increased alpha motor neuron excitability and increased H-reflex amplitude and following M-response, thus allowing measurement of the H-reflex, the M-response, and the H/M ratio

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of pysical therapy, MTI university, Cairo, Egypt